CLINICAL TRIAL: NCT00697970
Title: Study to Evaluate the Immunogenicity and Reactogenicity of Various Formulations of GSK Biologicals' (Previously SmithKline Beecham Biologicals') Recombinant Hepatitis B Vaccine in Healthy Adult Volunteers
Brief Title: Evaluation of Immunogenicity and Reactogenicity of Various Formulations of Recombinant Hepatitis B Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 208129/006
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Engerix™-B; Recombinant Hepatitis B vaccine; Adjuvant
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (6):
- Group A (Experimental)
  Interventions: Biological: HBsAg formulated with different concentrations of MPL and Aluminium Salts
- Group B (Experimental)
  Interventions: Biological: HBsAg formulated with different concentrations of MPL and Aluminium Salts
- Group C (Experimental)
  Interventions: Biological: HBsAg formulated with different concentrations of MPL and Aluminium Salts
- Group D (Experimental)
  Interventions: Biological: HBsAg formulated with different concentrations of MPL and Aluminium Salts
- Group E (Experimental)
  Interventions: Biological: HBsAg formulated with different concentrations of MPL and Aluminium Salts
- Group F (Active Comparator)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBsAg formulated with different concentrations of MPL and Aluminium Salts — Intramuscular injection, 3 doses
  Arms: Group A; Group B; Group C; Group D; Group E
Biological: Engerix™-B — Intramuscular injection, 3 doses
  Arms: Group F

SUMMARY:
The purpose of the present trial is to evaluate 6 vaccine formulations of recombinant hepatitis B vaccine for their reactogenicity and immunogenicity when administered at 0-2 months with a booster at month 12

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years old.
* Written informed consent will have been obtained from the subjects.
* Good physical condition as established by physical examination and history taking at the time of entry.
* Female participants will avoid becoming pregnant during the study period and they will have been on a contraceptive program for at least 2 months before entry.

Exclusion Criteria:

* Pregnancy or lactation.
* Positivity for anti hepatitis antibodies.
* Any vaccination against hepatitis B in the past.
* Any previous administration of MPL.
* Elevated serum liver enzymes.
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Axillary temperature > 37.5°C at the time of injection.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Any treatment with immunosuppressive or immunostimulant therapy.
* Any chronic drug treatment, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Administration of any other vaccine(s) or any immunoglobulin during the study period.
* Simultaneous participation in any other clinical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 321 (Actual)
Dates: Start 1993-11; Primary Completion 1995-04 (Actual); Study Completion 1995-04 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | After two doses and after the booster dose

SECONDARY OUTCOMES:
Occurrence and intensity of local and general solicited symptoms | 8 days after vaccination
Anti-HBs antibody concentrations | Screening, M1, 2, 3, 4, 6, 12, 13
Occurrence of unsolicited adverse events | 30-day after vaccination
Occurrence of serious adverse events | During the study period and 30 days after the last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Vienna, Austria